CLINICAL TRIAL: NCT01942629
Title: Prognostic Value of Quantitative p63 Immunostaining in Adenocarcinoma of Lung, Breast, and Pancreas
Brief Title: Prognostic Value of the Marker P63 in Adenocarcinoma of Lung, Breast, and Pancreas
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, SHOROOK NA'ARA MD, MD, Rambam Health Care Campus
Other Study IDs: 0298-13ctil
Record Dates: First submitted 2013-08-22; First posted 2013-09-16 (Estimated); Last update posted 2013-09-16 (Estimated); Status verified 2013-09

CONDITIONS: Lung Adenocarcinoma; Breast Adenocarcinoma; Pancreatic Ductal Adenocarcinoma
Keywords: prognostic markers,Pancreatic ductal adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma of Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Lung adenocarcinoma: This group will include 100 patients with lung adenocarcinoma, the clinical outcomes will be retrospectively assessed.
  at the same time 2 histopathological slides will be retrieved and stained for known markers as well as to P63.
  Interventions: Other: their will be no intervention in any of the groups, the study is retrospective
- Breast adenocarcinoma: This group will include 100 patients with breast adenocarcinoma, the clinical outcomes will be retrospectively assessed.
  at the same time 2 histopathological slides will be retrieved and stained for known markers as well as to P63.
  Interventions: Other: their will be no intervention in any of the groups, the study is retrospective
- Pancreatic ductal adenocarcinoma: This group will include 100 patients with pancreatic ductal adenocarcinoma, the clinical outcomes will be retrospectively assessed.
  at the same time 2 histopathological slides will be retrieved and stained for known markers as well as to P63.
  Interventions: Other: their will be no intervention in any of the groups, the study is retrospective

INTERVENTIONS:
Other: their will be no intervention in any of the groups, the study is retrospective

SUMMARY:
The p63 gene is a recently discovered member of the p53 family located at chromosome 3q27Many studies have reported that overexpression of p63 can mimic p53 activities by binding DNA, activating transcription, and inducing apoptosis.

Various studies proved p63 as a marker of basal cells in normal salivary glands, breast, prostate, respiratory and squamous epithelia, and of tumor cells from various malignancies. Still, p63 has been the subject of relatively few studies in lung adenocarcinoma, and breast carcinoma, and no study has described the correlation of p63 with pancreatic ductal adenocarcinoma.

In the current study, we aim to evaluate the prognostic value of the expression of p63 in the lung adenocarcinoma, breast adenocarcinoma, and pancreatic ductal adenocarcinoma. We will achieve this aim by collecting clinical data retrospectively from the patients' medical records as well as assessing the histological sections and performing immunohistochemical staining for p63.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were treated at our institution for lung adenocarcinoma, breast adenocarcinoma, or pancreatic ductal adenocarcinoma.
* Available histopathological diagnosis of the malignancy.

Exclusion Criteria:

* Patients with inoperable tumors.
* Patients with second primary tumor.
* Patients with pathological blocks not enough for future slicing.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 300 patients, 100 for each group.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-10 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
5 year overall survival | 5 years
  if the patient is alive or dead 5 years following the treatment

SECONDARY OUTCOMES:
recurrence free survival | 5 years
  the recurrence of the disease within 5 years from the treatment